CLINICAL TRIAL: NCT00131443
Title: A Double-Blind Dose Comparison Study of Topiramate in Pediatric Subjects With Basilar/Hemiplegic Migraine
Brief Title: Dose Comparison Study of Topiramate in Pediatric Subjects With Basilar/Hemiplegic Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Monarch Medical Research (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CAPSS 271
Record Dates: First submitted 2005-08-15; First posted 2005-08-18 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2006-11

CONDITIONS: Basilar Migraine
Keywords: Basilar/Hemiplegic Migraine; Prophylaxis
MeSH Terms: conditions — Migraine with Aura | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The objective of this study is to assess the effectiveness and safety of topiramate in the prevention of basilar and hemiplegic migraine in children and adolescents.

DETAILED DESCRIPTION:
The objective of this study is to assess the efficacy and safety of topiramate in the prophylaxis of basilar migraine and hemiplegic migraine in children and adolescents, by comparing two doses, 25 and 100 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Must meet International Headache Society (IHS) classification of pediatric migraine with aura: familial hemiplegic migraine (International Classification of Headache Disorders [ICHD] 1.2.4), sporadic hemiplegic migraine (ICHD 1.2.5) or basilar-type migraine (ICHD 1.2.6).
* Average of 4 migraine-days/month during the 3 months prior to screening.
* 4 migraine-days during prospective baseline period.
* At least one of the subject's migraines during the previous 3 months must have been accompanied by their characteristic basilar-type or hemiplegic neurologic symptoms of moderate to severe degree.
* 6-18 years of age.
* Weigh more than 25 kg.
* If female, subjects must:

  1. be premenarchal or otherwise incapable of pregnancy, or
  2. have practiced one of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, spousal/partner sterility, or
  3. be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence.

If (b) or (c), the subject must have a negative urine pregnancy test within one week of study entry.

* Able to take oral medication in tablet form
* Willing and able to:

  1. read and comprehend written instructions,
  2. complete the assessment forms,
  3. return for regular visits, and d) adhere to medication regimens.

Exclusion Criteria:

* Previously failed topiramate therapy for migraine prophylaxis or those who discontinued topiramate due to adverse events.
* Have taken topiramate within 14 days prior to the start of the prospective baseline period.
* Have 15 or more headache-days during the prospective baseline period.
* Have cluster headaches or chronic migraine.
* Have migraine aura without headache exclusively.
* Currently have a more painful condition than their migraine pain.
* Have taken any medications for migraine prophylaxis, within 2 weeks of the start of the prospective baseline period.
* Progressive neurological disorders or a structural disorder of the brain
* Overuse analgesic or migraine-specific agents for abortive treatment of migraine:

  * >10 treatment days/month of ergot-containing medication, triptans, or opioids;
  * >15 treatment days/month with simple analgesics (including NSAIDs)
* Require any injections of corticosteroids or local anesthetics within 60 days of visit 1 or botulinum toxin within 120 days prior to Visit 1.
* Have previously failed more than 2 adequate trials of an established prophylactic anti-migraine regimen.
* Subjects starting non-pharmacologic prophylactic approaches within 1 month prior to Visit 1. Non-pharmacologic prophylactic approaches started at least 1 month prior to Visit 1 should be continued throughout the study.
* Have taken carbonic anhydrase inhibitors or triamterene within 1 month prior to Visit 1.
* History of nephrolithiasis.
* Require continuing treatment with anticonvulsant therapy for a non-migraine condition.
* Significant major psychiatric disorder (e.g., major depression) or subjects receiving anti-psychotic medication.
* History of attempted suicide or suicidal tendencies.
* History of substance abuse.
* Pregnant or lactating females.
* Clinically unstable neurological, cardiovascular, gastrointestinal, musculoskeletal, pulmonary or other disease.
* Active liver disease.
* AST and/or ALT levels greater than 2 times the upper limit of normal range.
* Received an investigational drug or used an investigational device within 30 days of study entry.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2006-08

PRIMARY OUTCOMES:
The primary efficacy outcome will be the reduction in average monthly migraine-days over the entire double-blind phase relative to the prospective baseline period

SECONDARY OUTCOMES:
Reduction in frequency, severity and duration of basilar or hemiplegic aura symptoms
Reduction in migraine pain severity and duration
Reduction in migraine episode and headache episode frequency
Reduction in total headache days
Proportion of responders (i.e., the proportion of subjects who experience a ≥ 50% reduction in migraine-days and migraine episodes)
Cumulative reduction in frequency of migraine days and migraine episodes
Reduction in the use of acute/abortive medications
Reduction in migraine-associated symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Lewis, MD, Principal Investigator — Monarch Medical Research
Locations (1):
- Monarch Medical Research - Child and Adolescent Neurology, Norfolk, Virginia, United States